CLINICAL TRIAL: NCT04474717
Title: Clinical and Biochemical Assessment of the Course of Chronic Obstructive Pulmonary Disease in Combination With Atherosclerosis
Brief Title: Chronic Obstructive Pulmonary Disease in Combination With Atherosclerosis (Clinical and Biochemical Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 15.06.2020
Record Dates: First submitted 2020-06-29; First posted 2020-07-17 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2021-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Peripheral Artery Disease
Keywords: COPD; peripheral atherosclerosis; comorbidity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Peripheral Arterial Disease | interventions — Physical Examination; Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The natural history of COPD (Other): Monitoring risk factors, chronic respiratory symptoms and respiratory function in the natural history of chronic obstructive pulmonary disease
  Interventions: Diagnostic Test: clinical examination, spirometry
- Study of systemic inflammation and molecular mechanisms (Experimental): Study of systemic inflammation and molecular mechanisms underlying the comorbid course of COPD and atherosclerosis
  Interventions: Diagnostic Test: blood monocyte assay
- Exhaled breath condensate (Other): A study of the clinical and biochemical COPD phenotype with systemic inflammation and comorbidity
  Interventions: Diagnostic Test: Breath Condensate Collection

INTERVENTIONS:
Diagnostic Test: Breath Condensate Collection — Breath Condensate Collection
  Arms: Exhaled breath condensate
Diagnostic Test: clinical examination, spirometry — spirometry
  Arms: The natural history of COPD
Diagnostic Test: blood monocyte assay — study of blood monocytes in the laboratory of cell technology
  Arms: Study of systemic inflammation and molecular mechanisms

SUMMARY:
one-centered, open, non-randomized, controlled clinical trial will focus on a comprehensive study of the clinical, functional and molecular biochemical characteristics of the natural course of COPD in combination with peripheral atherosclerosis

DETAILED DESCRIPTION:
Risk factors, chronic respiratory symptoms and respiratory function in the natural history of COPD will be monitored. In a group of patients with a comorbid course of COPD and atherosclerosis, systemic inflammation and its molecular mechanisms will be investigated. Also in this group, the role of non-coding miRNAs will be analyzed. The study also includes an analysis of the clinical and biochemical COPD phenotype with systemic inflammation and comorbidity.

ELIGIBILITY:
Inclusion Criteria:

1. A significant diagnosis of COPD, confirmed by spirometry criteria, typical clinical presentation.
2. A significant diagnosis of peripheral atherosclerosis
3. The high level of adherence to treatment
4. Signed informed agreement

Exclusion Criteria:

1. The presence of other chronic respiratory diseases in the patient, including bronchial asthma
2. Known oncological diseases of any localization
3. HIV infection and other immunodeficiency conditions
4. Inability to understand and comply with the requirements of the research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
mortality | 12 months
  the number of deaths from cardiovascular causes
lung function | 12 months
  progression of decreased lung function (FEV1%) according to spirometry
exacerbations | 12 months
  frequency of exacerbations of COPD (number of cases per year)
markers of inflammation | 12 months
  biochemical markers of inflammation (IL-6, pg/ml; IL-8,pg/ml;TNF,pg/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Ryazan State Medical University, Ryazan, Please Select, Russia

IPD SHARING:
Plan to Share IPD: No